CLINICAL TRIAL: NCT03411603
Title: Food and Diet Based Validations of a Nutrient Profiling System for Reformulation in Two Nationally Representative Surveys
Brief Title: Validation of a Nutrient Profiling System for Reformulation
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: AJCN/2017/172213
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Nutrition Poor
Keywords: nutrient profiling
MeSH Terms: conditions — Malnutrition | interventions — Diet

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- INCA2 2006-07: French National Dietary Intake Survey, conducted in 2006-2007 by the French Agency for Food, Environmental and Occupational Health Safety.
  Adults aged 18y and over, n=1918 included in the analyses.
  Interventions: Other: Diet and socio-demographic questionnaires
- NHANES 2011-12: Wave 2011-12 of the National Health and Nutrition Examination Survey, the US national dietary intake Survey, conducted by the Centers for Disease Control and Prevention (CDC) Adults aged 18y and over, n=5073 included in the analyses.
  Interventions: Other: Diet and socio-demographic questionnaires

INTERVENTIONS:
Other: Diet and socio-demographic questionnaires — 24-hr recall or food diary questionnaires; socio-demographic questionnaires

SUMMARY:
The objectives of the study are to assess the validity of Nestlé reformulation criteria in two national dietary surveys: the US NHANES 2011, and the French INCA2 2006-07.

DETAILED DESCRIPTION:
Background: The Nestlé Nutritional Profiling System (NNPS) has been developed to guide food and beverage reformulation. It is not known whether products passing the NNPS standards have a higher overall nutritional density, and whether the higher consumption of NNPS Pass products is associated with a higher dietary quality.

Objective: The objectives were (i) to compare the classifications derived from the NNPS and the validated UK Ofcom nutrient profiling system; and (ii) to assess the NNPS construct validity against healthy and unhealthy diets in French (Individual and National Survey on food Consumption 2006-2007) and the US (National Health and Nutrition Examination Surveys 2011-2012) nationally representative dietary surveys.

Design: NNPS outcomes (PASS, FAIL, Out-of-scope) of foods were compared to UK Ofcom outcomes. Contributions of NNPS outcomes to energy intakes were compared between diets nutritional quality classes defined by two methods: based on a food-based quality indicator (PNNS-GS in France, HEI-2010 in the US), or on a combination of three nutrient-based indicators (MAR, MER, energy density).

ELIGIBILITY:
Inclusion Criteria:

* All participants of INCA2 and NHANES 2011-12 surveys

Exclusion Criteria:

* Missing dietary intake data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative samples of the US and French adult populations
Sampling Method: Probability Sample
Enrollment: 6991 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Index 2010 | 2011-12
  Measure of dietary quality for the NHANES Survey, based on reported dietary intakes
PNNS-GS diet score | 2006-07
  Measure of dietary quality for the French INCA2 Survey, based on reported dietary intakes

SECONDARY OUTCOMES:
Mean Adequacy Ratio | 2006-07 and 2011-12
  Measure of individuals nutrient adequacy based on reported food intakes
Mean Excess Ratio | 2006-07 and 2011-12
  Measure of excessive nutrient consumption, based on reported food intakes
Energy density | 2006-07 and 2011-12
  Solid energy density of diets, based on reported food intakes

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Porter, Study Director — Centers for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No
The NHANES 2011-12 and INCA2 data are available to other researchers via the respective websites.

REFERENCES:
- See also: Details of French dietary surveys. ANSES website — https://www.anses.fr/en/content/inca-studies